CLINICAL TRIAL: NCT04539782
Title: A Feasibility Study on the Value of Pelvic Floor Training After Pelvic Organ Prolapse Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Landspitali University Hospital (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LSH-20-001
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic floor; physiotherapy; pelvic organ prolapse; post op; recurrence
MeSH Terms: conditions — Pelvic Organ Prolapse; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy intervention (Experimental): Pelvic floor muscle training given by a physiotherapist in four sessions and follow up phone calls twice in 14 weeks
  Interventions: Other: Physiotherapy intervention
- No intervention (No Intervention): Standard care

INTERVENTIONS:
Other: Physiotherapy intervention — Compare the effect of structured pelvic floor muscle training supported by physiotherapist post operation on POP on recurrence of symptoms or symptoms in a new compartment, quality of life and pelvic floor muscle function.
  Arms: Physiotherapy intervention

SUMMARY:
The main objective is to assess the feasibility of a randomized controlled trial that investigates the effects of pelvic floor training on recurrence in pelvic organ prolapse surgeries. This will be achieved by measuring POP-Q stage and by a validated questionnaire before surgery and one year after. Women having POP surgery at Landspitali will be offered to participate if they meet the criteria of the research. Participants will be randomized into two groups, interventions and control group that gets standard care at the hospital. The intervention group will meet a physiotherapist 6 weeks post-op for targeted physiotherapy with pelvic floor training, conventional advice and support. Over 16 weeks period participants in intervention group will get physiotherapy four times and get two follow up phone calls. Pelvic floor activity will be measured with EMG and symptoms collected with questionnaire before surgery and year post-op.

Recurrent surgeries are common problem shortly after the first one. POP symtoms can be bothersome for women and reduce their quality of life. More knowledge is needed to figure out if targeted physiotherapy with pelvic floor training can help reduce recurrency and bothersome symptoms.

DETAILED DESCRIPTION:
A feasibility study to assess the practicality of physiotherapy treatment after pelvic organ prolapse (POP) surgery and the effect on recurrent POP symptoms, pelvic floor activity and general physical fitness.

Pelvic organ prolapse is a common problem among women and many do need surgery. Little is known about recurrence of POP surgeries. Pelvic floor muscle training (PFMT) has positive effects on POP symptoms and quality of life. Research shows PFMT can reduce stage of the prolapse.

Before surgery POP-Q stage will be measured by urogynocologist. Pelvic floor muscle activity will be measured with EMG vaginal probes. General physical fitness will be tested with 30s chair-stand and core strenght with prone bride test. An Icelandic version of The Australian Female PelvicFloor questionnaire will be used to assess symptoms and affect on quality of life.

Participants will be randomized into two groups, intervention and control group. The control group gets standard care at the hospital. The interventional group gets physiotherapy with PFMT, conventional advise and support. During 16 weeks intervention participants get four sessions with specialized physiotherapist and two follow up phone calls. Follow up measures will be made at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women having their first POP surgery at LSH
* <80 years old
* Icelandic speaking

Exclusion Criteria:

* Women that previously have had incontinence surgery, hysterectomy or previous POP surgery.
* Dementia, physical disabilities that could affect the research, previous radiotherapy and neurological diseases.
* Women participating in the research that need to have recurrent POP surgery or incontinence surgery within the year of the surgery.

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
POP-Q | One year
  POP-Q stages are measured by urogynocologists who are blinded outcome assessors.

SECONDARY OUTCOMES:
The Australian Female Pelvic Floor Questionnaire | One year
  Pelvic floor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Þorgerður Sigurðardóttir, MSc, Principal Investigator — Landspítali University Hospital/University of Iceland, Reykjavík, Iceland.; Helga Medek, MD, MSc, Study Chair — Landspítali University Hospital/University of Iceland, Reykjavík, Iceland.; Þórarinn Sveinsson, PhD, Study Chair — University of Iceland
Locations (1):
- Landspitali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No